CLINICAL TRIAL: NCT06541340
Title: A New Strategy for Preoperative Drainage of Resectable Pancreatic Head Cancer Combined Severe Obstructive Jaundice, a Multicenter, Open-label, Randomized Controlled Clinical Study
Brief Title: A New Strategy for Preoperative Drainage of Resectable Pancreatic Head Cancer Combined Severe Obstructive Jaundice
Acronym: PROB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROB
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer; Obstructive Jaundice
Keywords: pancreatic head cancer; obstructive Jaundice; preoperative biliary drainage; prealbumin
MeSH Terms: conditions — Pancreatic Neoplasms; Jaundice, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional strategy (Active Comparator): Traditional preoperative biliary drainage strategy with total bilirubin as the main indicator
  Interventions: Procedure: Traditional strategy
- Modified strategy (Experimental): Modified preoperative biliary drainage strategy with prealbumin as the main indicator
  Interventions: Procedure: Modified strategy

INTERVENTIONS:
Procedure: Modified strategy — Modified preoperative biliary drainage strategy with prealbumin as the main indicator
  Arms: Modified strategy
Procedure: Traditional strategy — Traditional preoperative biliary drainage strategy with total bilirubin as the main indicator
  Arms: Traditional strategy

SUMMARY:
Severe obstructive jaundice caused by pancreatic head cancer usually requires preoperative biliary drainage, but its necessity and effectiveness are controversial, and specific strategies lack clear standards. This study proposed a new strategy for preoperative biliary drainage using serum prealbumin as the main evaluation index, and compared it with the traditional strategy using serum total bilirubin as the main evaluation index. Through a randomized, controlled, multicenter prospective study, we explored the effects of different drainage strategies on the incidence of in-hospital complications and long-term prognosis of patients with resectable pancreatic head cancer, guided clinical decisions on preoperative drainage time and surgical timing, and provided high-quality evidence-based medicine for preoperative biliary drainage of pancreatic head cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of pancreatic head cancer, or clinical diagnosis of pancreatic head cancer after multidisciplinary discussion, clear presence of obstructive jaundice caused by pancreatic head tumor, and planned to undergo radical pancreaticoduodenectomy
2. Preoperative imaging stage is resectable
3. Baseline serum total bilirubin ≥ 250μmol/L, and no history of preoperative biliary drainage
4. Age >18 and ≤75 years old
5. ECOG(Eastern Cooperative Oncology Group) physical score ≤ 2
6. Signed informed consent, received preoperative endoscopic biliary drainage (ERCP) and radical surgery timing evaluation

Exclusion Criteria:

1. Combined with other malignant tumors
2. Combined with uncontrolled medical diseases or organ dysfunction and other absolute counterindications for surgery
3. Pregnant and lactating women
4. Patients who cannot tolerate preoperative biliary drainage or radical surgery
5. Other situations that are not suitable for inclusion in clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital complications | During hospitalization, up tp 3 months
  In-hospital complications are comprehensively evaluated by the chief surgeon, responsible doctor and their team based on clinical manifestations, laboratory tests, etc., and reviewed by the expert committee of this study. The name of the complication, time of occurrence, treatment measures and outcome are strictly recorded.

SECONDARY OUTCOMES:
Recurrence/metastasis | 12 months after discharge
  It is mainly based on follow-up. If the follow-up was completed in our hospital, the hospital system will be directly retrieved to obtain the diagnosis information. The follow-up was conducted by interviewing the patient or his family members through telephone questionnaires or face-to-face visits to collect required information.The follow-up subjects provide medical records, etc., and record in detail the time of diagnosis of long-term complications or recurrence and metastasis, diagnostic basis, laboratory tests, treatment measures and outcomes, which must be reviewed by the expert committee of this study.
Mortality | 12 months after discharge
  It is mainly based on follow-up. If the follow-up was completed in our hospital, the hospital system will be directly retrieved to obtain the diagnosis information. The follow-up was conducted by interviewing the patient or his family members through telephone questionnaires or face-to-face visits to collect required information.The follow-up subjects provide medical records, etc., and record in detail the time of diagnosis of long-term complications or recurrence and metastasis, diagnostic basis, laboratory tests, treatment measures and outcomes, which must be reviewed by the expert committee of this study.
Long-term complications | 12 months after discharge
  It is mainly based on follow-up. If the follow-up was completed in our hospital, the hospital system will be directly retrieved to obtain the diagnosis information. The follow-up was conducted by interviewing the patient or his family members through telephone questionnaires or face-to-face visits to collect required information.The follow-up subjects provide medical records, etc., and record in detail the time of diagnosis of long-term complications or recurrence and metastasis, diagnostic basis, laboratory tests, treatment measures and outcomes, which must be reviewed by the expert committee of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No